CLINICAL TRIAL: NCT05968586
Title: Effect of Body Position on Oxygenation, Ventilation, and Diaphragmatic Workload in Premature Infants on Non-Invasive Neurally Adjusted Ventilatory Assist (NAVA)
Brief Title: Non-Invasive Neurally Adjusted Ventilatory Assist (NAVA) Prone vs Supine in Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Nada Darwish, Neonatal-Perinatal Medicine Fellow, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22600
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Neonatal Oxygen Desaturation; Premature; Ventilator Lung; Newborn; Apnea of Prematurity
Keywords: apnea of prematurity; NAVA
MeSH Terms: conditions — Asphyxia Neonatorum; Premature Birth; Bronchopulmonary Dysplasia; Apnea | interventions — Posture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prone positioning (Experimental)
  Interventions: Other: Body positioning
- Supine positioning (Active Comparator)
  Interventions: Other: Body positioning

INTERVENTIONS:
Other: Body positioning — Body positioning of infants prone vs supine.

SUMMARY:
This research study is being done to investigate the effect of changing an infant's body position on how hard the baby works to breathe, the baby's oxygen level, the baby's carbon dioxide level, the baby's lung volume, the baby's lung compliance (ability of the lung to expand and fill with air), and how frequently the baby develops clinically significant events such as apnea (baby stops breathing on his own), bradycardia (low heart rate), and desaturation (low oxygen) events.

ELIGIBILITY:
Inclusion Criteria:

* Viable infants born at ≤32 weeks of gestation on non-invasive NAVA.
* Infant must be stable on NAVA for at least 24 hours prior to the study

Exclusion Criteria:

* Infants with congenital heart disease (CHD)
* Infants with persistent pulmonary hypertension (PPHN)
* Infants with contraindications to using NAVA (e.g. neuromuscular blockage or paralysis, absent electrical signal from the diaphragm, esophageal tears or bleeding, cardiac pacemakers) or infants in whom an NG/OG catheter cannot be placed.

Ages: 1 Minute to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-12-28 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Peak electrical activity of the diaphragm (Edi peaks) | From enrollment in study to end of study (a total of twelve hours)
  Height of Edi signal in uV
Minimum electrical activity of the diaphragm (Edi mins) | From enrollment in study to end of study (a total of twelve hours)
  Lowest of Edi signal in uV
Number of apenic events | From enrollment in study to end of study (a total of twelve hours)
  Number of times where infant ceases to breath for >5 seconds
Number of bradycardia events | From enrollment in study to end of study (a total of twelve hours)
  Number of times where infant's heart rate drops <100bpm sustained for >5s
Number of desaturation events | From enrollment in study to end of study (a total of twelve hours)
  Number of times where infant's oxygen saturation drops <85% sustained for >5s

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Glass, MD, Study Director — Penn State College of Medicine
Locations (1):
- Penn State Health Milton S Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No